CLINICAL TRIAL: NCT01626144
Title: Metabolizing Enzyme Genotype Versus Exemestane Metabolism Profiles
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 35099EP
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: Exemestane; Metabolism; Metabolizing enzyme genotype; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer, exemestane treatment: Breast cancer patients receiving standard of care exemestane

SUMMARY:
It is the investigators hypothesis that exemestane (EXE) metabolism is an important source of the inter-individual variation in EXE metabolic profiles and that polymorphisms in EXE-metabolizing enzymes may potentially play a role in affecting EXE therapeutic efficacy and toxicity. The goals of this clinical study are to (1) establish EXE metabolism profile kinetics, and (2) determine whether correlations exist in vivo between metabolizing enzyme genotype and urinary EXE metabolite profiles in women being treated with EXE. Together, these studies will allow us to fully characterize functionally-relevant polymorphisms in the EXE-metabolizing enzyme pathway that are potentially important in EXE clinical efficacy.

DETAILED DESCRIPTION:
Aromatase inhibitors (AIs) are widely used as adjuvant treatment for estrogen-receptor positive breast cancer in post-menopausal women. AIs have been demonstrated to have equal to or greater efficacy and less toxicity than tamoxifen (TAM), the drug of choice for many years. Exemestane (EXE) is a 3rd-generation AI that has demonstrated efficacy in the treatment of breast cancer patients, and as with TAM and other AIs, there has been considerable inter-individual variability in overall response to EXE and in the occurrence of toxicities, but the causes of this variability have not been elucidated. Differences in drug metabolism can be a source of variability between patients. Genetic variations occur in several of the enzymes involved in phase I and II metabolic reactions and many of these can lead to alterations in enzyme activity which in turn can alter therapeutic response to drugs. EXE is extensively metabolized as unchanged EXE and is found at less than 1% in urine and 10% in plasma. EXE pharmacokinetics will be established in a series of 20 subjects taking EXE. EXE metabolites will then be measured at an optimal time post-EXE dose in the urine of 200 breast cancer patients being treated with EXE to establish whether metabolizing enzyme genotype-EXE metabolism phenotype correlations exist in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who have ER+ tumors and are taking 25 mg EXE daily (orally)
* Post-menopausal women or chemically post-menopausal women (who won't become pregnant since they are taking zoladex), or women who are post-menopausal as a result of ovary removal
* Patients may be at any point in their hormonal treatment, but must have completed any planned surgery, radiation and chemotherapy.

Exclusion Criteria:

* Concurrent use of corticosteroids, megestrol, or phenobarbitol (inhaled and internasal steroids are permitted)
* History of allergy to exemestane

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal breast cancer patients in the breast oncology clinic at the Penn State Hershey Cancer Institute (PSHCI).
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Metabolizing enzyme genotype vs EXE metabolism profiles | 6 years
  Functional genotypes will be determined for EXE-metabolizing enzymes and will be correlated with blood/urinary EXE metabolism profiles

SECONDARY OUTCOMES:
EXE toxicities | 6 years
  Patient-reported EXE-induced toxicities will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lazarus, Ph.D., Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States